CLINICAL TRIAL: NCT01959568
Title: Double Endotamponade With Perfluorodecalin and Silicone Oil in Retinal Detachment Surgery: Randomised Clinical Trial of Safety
Brief Title: Double Endotamponade With Perfluorodecalin and Silicone Oil in Retinal Detachment Surgery.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The S.N. Fyodorov Eye Microsurgery State Institution (Other Government)
Responsible Party: Principal Investigator, Pavel V. Lyskin, Pavel V. Lyskin, MD, PhD, The S.N. Fyodorov Eye Microsurgery State Institution
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: #8, 04/09/2013
Record Dates: First submitted 2013-09-29; First posted 2013-10-10 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2014-05

CONDITIONS: Retinal Detachment
Keywords: Retinal Detachment; Double Tamponade; Perfluorocarbon liquids; Vitrectomy
MeSH Terms: conditions — Retinal Detachment | interventions — Vitrectomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Double tamponade (Experimental): Vitrectomy and tamponade: subtotal vitrectomy, epiretinal membrane removal, perfluorodecalin tamponade, retinal photocoagulation. After that the surgeon replaces ½ of perfluorodecalin volume by silicone oil.
  Interventions: Procedure: Vitrectomy and tamponade
- Silicone oil tamponade (Active Comparator): Vitrectomy and tamponade: subtotal vitrectomy, epiretinal membrane removal, perfluorodecalin tamponade, retinal photocoagulation and perfluorodecalin-silicone oil exchange.
  Interventions: Procedure: Vitrectomy and tamponade

INTERVENTIONS:
Procedure: Vitrectomy and tamponade — In the double tamponade arm the result of surgery is vitreous cavity filled in a half with perfluorodecalin and in another half - with silicone oil.
  In the silicone oil tamponade arm the result of surgery is vitreous cavity filled with "conventional" or heavy silicone oil, depending on predominant retinal breaks location.
  Other Names: Perfluorodecalin Dk-Line (Bausch&Lomb); Silicone oil Oxane 1300 (Bausch&Lomb); Silicone oil Oxane HD (Bausch&Lomb)

SUMMARY:
Purpose: to assess the efficacy and safety of double tamponade versus silicone oil tamponade.

Design: parallel-group study with balanced [1:1] stratified block randomization. Eligible participants are all adults aged 18 or over with first diagnosed rhegmatogenous total retinal detachment with retinal breaks located both in upper and lower retina. Also investigators include those patients with total retinal detachment with proliferative vitreoretinopathy (PVR) in which it is impossible to remove epiretinal membranes completely during the surgery (with arbitrary retinal breaks localization). Exclusion criteria are severe concomitant eye pathologies (glaucoma, diabetic retinopathy, macular hole, traumas etc) and eye length more than 27mm.

Patients are randomized in two groups (test group and control group).

In the test group patients undergo subtotal vitrectomy, epiretinal membrane removal, perfluorodecalin (PFD) tamponade, retinal photocoagulation. After that the surgeon replaces ½ of PFD volume by "conventional" SO (with density less than one of water). The result is vitreous cavity (VC) filled in a half with PFD and in another half - with SO. In the control group patients undergo subtotal vitrectomy, epiretinal membrane removal, PFD tamponade, retinal photocoagulation and PFD-SO exchange, so the result is VC filled with "conventional" or heavy SO, depending on predominant retinal breaks location. 30 days after the surgery in both groups tamponing agents are removed from VC and VC is filled with sulfur hexafluoride gas (SF6) which dissolves during 1 month. Follow-up is at least 12 months.

Along with standard examinations, after SF6 gas dissolution investigators perform spectral optical coherence tomography (OCT) and microperimetry. With OCT investigators measure thickness of retinal inner and outer nuclear layers. With microperimetry investigators determine light sensitivity in 12° and 4° zones from the fixation point.

Outcome measures: reattachment rate, best corrected visual acuity (BCVA), intraocular pressure (IOP), thicknesses of inner and outer nuclear layers according to the OCT, light sensitivity according to microperimetry, the rate of cataract formation in phakic eyes and the rate of tamponing agents emulsification.

For final analysis each group will include 145 participants.

OCT, microperimetry data and visual acuity will be compared between the groups using Student's t-test; proportions will be compared using exact Fisher's test.

DETAILED DESCRIPTION:
The investigators include in the study all successive patients operated by the same surgeon. The study takes place in the S.N. Fyodorov "Eye Microsurgery" Federal State Institution located in Moscow, Russian Federation.

Patients are randomized in two groups with stratified block randomization. Strata were defined by combination of two binary prognostic factors: duration of retinal detachment (less than 3 months and ≥ 3 months) and PVR (present/absent).

Early interim analysis will be performed in order to reveal possible adverse effect of long-term PFD tamponade. For interim report success will mean the rate of post-surgical BCVA >/= 20.200. Groups sizes for interim analysis will be 35 patients in each group. For interim analysis the investigators choose group sizes able to reveal 30% absolute difference in functional success rate with one-sided test (to detect possible toxicity of double tamponade for the retina) having power of 0.8 and significance level of p=0.05. In the final analysis success will mean retinal reattachment.

For final analysis each group will include 145 participants, so that the investigators are able to detect 15% difference in reattachment rate with power of 0.8 and significance level of p=0.05. Group sizes were computed with exact Fisher's test function in G*Power 3.1.7 software (Erdfelder, Faul, & Buchner).

OCT is performed with Cirrus HD-OCT system (Zeiss Meditec Inc). Microperimetry is performed with MP-1 microperimeter (Nidek). All the examinations are assessed by one ophthalmologist.

The allocation concealment is implemented with the help of a third party, who stores the randomization list and prepares envelopes containing directions what method of tamponade to employ in each particular patient. Patients are blind to the method of tamponade.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 18 or over with firstly diagnosed rhegmatogenous total retinal detachment:

1. with retinal breaks located both in upper and lower retina; OR
2. with PVR which was impossible to remove completely during the surgery.

Exclusion Criteria:

1. severe concomitant eye pathologies (glaucoma, diabetic retinopathy, macular hole, traumas); OR
2. eye length more than 27mm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2010-03; Primary Completion 2017-09 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Retinal reattachment rate | in 1 month after tamponade removal.

SECONDARY OUTCOMES:
Percentage of patients with best corrected visual acuity >/= 20.200 | in 1 month after tamponade removal

OTHER OUTCOMES:
Percentage of patients with intraocular pressure >/= 25 mm Hg | in 1 month after tamponade removal.
Percentage of phakic eyes in which cataract occurred during tamponade | During tamponade removal.
Percentage of eyes with tamponing substances emulsification | During tamponade removal.
Thickness of retinal inner and outer nuclear layers | in 1 month after tamponade removal
  Measured with Optical Coherence Tomography
Retinal light sensitivity | in 1 month after tamponade removal
  Measured with microperimetry

CONTACTS AND LOCATIONS:
Overall Officials: Pavel V Lyskin, PhD, Principal Investigator — SN Fyodorov "Eye Microsurgery" State Institution; Valery D Zakharov, Professor, Study Director — SN Fyodorov "Eye Microsurgery" State Institution
Locations (1):
- SN Fyodorov "Eye Microsurgery" State Institution, Moscow, Russia

REFERENCES:
- [Derived] Schwartz SG, Flynn HW Jr, Wang X, Kuriyan AE, Abariga SA, Lee WH. Tamponade in surgery for retinal detachment associated with proliferative vitreoretinopathy. Cochrane Database Syst Rev. 2020 May 13;5(5):CD006126. doi: 10.1002/14651858.CD006126.pub4. PMID 32408387